CLINICAL TRIAL: NCT04792515
Title: A Single-arm, Multicenter Clinical Study of Evaluating Camrelizumab Combined With SOX and/or Apatinib in the Treatment of Locally Advanced Gastric Cancer or Gastroesophageal Junction Adenocarcinoma
Brief Title: Camrelizumab Combined With SOX and/or Apatinib for Locally Advanced Gastric Cancer
Acronym: CCWSA/OAFLAG
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XJTU1AFCT-2021-003
Record Dates: First submitted 2021-03-07; First posted 2021-03-11 (Actual); Last update posted 2021-03-11 (Actual); Status verified 2021-01

CONDITIONS: Locally Advanced Gastric Cancer
Keywords: Camrelizumab ,Efficacy ,Safety
MeSH Terms: interventions — apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment group (Experimental): Patients were treated with camrelizumab combined with SOX/ or apatinib
  Interventions: Drug: Camrelizumab combined with SOX/ or apatinib

INTERVENTIONS:
Drug: Camrelizumab combined with SOX/ or apatinib — Camrelizumab: every 3 weeks (21 days) was given as one administration cycle. 200mg was given intravenously on the first day of each cycle. Dose adjustment is not allowed. Delayed administration is allowed.
  Apatinib mesylate: 250mg, qd, stopped 28 days before surgery, and can be used by the investigator according to the patient's recovery 28 days after surgery.
  Chemotherapy: The SOX regimen consisted of one cycle every 3 weeks (21 days).Dose adjustment is allowed. Delayed administration is allowed.
  Oxaliplatin (OXA) : 130mg/m2, intravenous infusion, d1, infusion more than 2 hours.
  Tigio Capsules (S-1) : Take orally after breakfast and dinner, twice daily, d1-14.
  The dosing time window is ±3 days, but within 72 hours before each dosing, subjects must complete an examination that includes all clinical requirements to assess tolerance for continued dosing.

SUMMARY:
This study was designed to evaluate the efficacy and safety of camrelizumab in combination with SOX and/or apatinib in the treatment of locally advanced gastric cancer or gastroesophageal junction adenocarcinoma.The primary endpoint was pathologic complete response (PCR).In addition, secondary efficacy endpoints include R0 resection rate, objective response rate (ORR), and 1-year progression-free survival rate (PFSR) . They were set to demonstrate the therapeutic benefit of camrelizumab combined with SOX in patients 。

DETAILED DESCRIPTION:
Screening period Subjects will enter the study screening period after signing the informed consent, and the maximum screening period will be 28 days. Those who meet all the inclusion criteria and do not meet the exclusion criteria will be allowed to enter the study treatment period.

Treatment period Patients received 2-4 cycles of neoadjuvant chemotherapy with camrelizumab +SOX regimen, and then received adjuvant chemotherapy with camrelizumab +SOX regimen after surgery, with a total of 8 cycles before and after surgery.

Camrelizumab: every 3 weeks (21 days) was given as one administration cycle. 200mg was given intravenously on the first day of each cycle. Dose adjustment is not allowed. Delayed administration is allowed.

Apatinib mesylate: 250mg, qd, stopped 28 days before surgery, and can be used by the investigator according to the patient's recovery 28 days after surgery.

Chemotherapy: The SOX regimen consisted of one cycle every 3 weeks (21 days).Dose adjustment is allowed. Delayed administration is allowed.

Oxaliplatin (OXA) : 130mg/m2, intravenous infusion, d1, infusion more than 2 hours.

Tigio Capsules (S-1) : Take orally after breakfast and dinner, twice daily, d1-14.

The dosing time window is ±3 days, but within 72 hours before each dosing, subjects must complete an examination that includes all clinical requirements to assess tolerance for continued dosing.

Subjects will continue to receive study therapy until disease progression (PD) occurs, intolerable toxicity occurs, a new antitumor therapy is initiated, treatment is terminated after careful consideration by the patient or investigator, or they die, or are lost to follow-up.

Clinical tumor evaluation during the screening period and throughout the study period will be based on RECIST version 1.1.Baseline tumor assessment was performed 28 days prior to the start of treatment.Enhanced computed tomography (CT) or magnetic resonance imaging (MRI) is recommended for tumor evaluation.Tumor efficacy evaluation was conducted every 2 cycles (±3 days) from the beginning of the first dose study until the occurrence of PD. The visit time for efficacy evaluation was fixed, regardless of whether the treatment cycle delay occurred.If treatment is discontinued for reasons other than PD, subjects will continue to undergo tumor evaluation until PD occurs, initiation of new antitumor therapy, withdrawal of informed consent, death, or loss of follow-up, whichever occurs first.In the event of clinical symptoms suggestive of PD, imaging methods should be used for subsequent evaluation in order to record and confirm tumor efficacy.

From the beginning of the first dose study treatment, a systematic safety assessment was carried out for each administration cycle.During the study treatment, a basic safety assessment was performed before each administration cycle, including completion of a physical examination, vital signs, and basic laboratory tests (ECG, blood routine, urine routine, fecal occult blood, blood biochemistry, coagulation function, etc.).

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign written informed consent before screening;
2. Male or female, ≥18 years old;
3. Have at least one measurable lesion according to RECIST1.1;
4. ECOG physical status score 0~1;
5. Pathologically confirmed local progression (CT3/CT4N+M0) of gastric cancer or adenocarcinoma of the gastroesophageal junction without any previous treatment (Siewert II or III).
6. According to the clinical staging standard, surgical treatment is planned after neoadjuvant chemotherapy.
7. Expected survival of more than 3 months;
8. The main organs function normally, following criteria:

I. Blood routine (no blood transfusion, no use of granulocyte colony stimulating factor (G-CSF) or other hematopoietic stimulating factor correction within 14 days before screening examination) : neutrophils ≥1.5× 109 /L, platelets ≥100×109/L, hemoglobin ≥90g/L;White blood cells acuity 3.5 x l09 / L II. Liver function: ALT and AST, ALT and AST ≤ 2.5×ULN; Total bilirubin (TBil) ≤ 1.5×ULN (Gilbert syndrome patients, ≤ 3×ULN); III. Renal function: serum creatinine (CR) ≤ 1.5×ULN or creatinine clearance (CCR) ≥60mL/ min; IV. Coagulation function: APTT, INR, PT ≤ 1.5×ULN;

Exclusion Criteria:

1. Gastric squamous cell carcinoma, adenosquamous cell carcinoma, small cell carcinoma and undifferentiated gastric carcinoma confirmed by pathology;
2. Positive HER-2 test (IHC3+ or IHC2+ amplified by FISH);
3. Any previous anti-tumor therapy (including chemotherapy, radiotherapy, hormone therapy, and molecular targeted therapy);
4. Cardiac and pyloric obstruction affects the patient's eating and gastric emptyor and has difficulties to swallow tablets;
5. Previous immunotherapy with anti PD-1, anti PD-L1, anti PD-L2, anti CD137 or anti CTLA-4 antibodies or any other antibodies or drugs that target co-stimulation of T cells or immune checkpoint pathways;
6. Has developed or is currently having other malignant tumors within 5 years, except for cured cervical carcinoma in situ, non-melanoma skin cancer, or other tumors/cancers that have undergone radical treatment and have been free of disease for at least 5 years;
7. Perimeter neuropathy is grade 2 or greater according to the common adverse event terminology (NCI-CTCAE V5.0);
8. with known active central nervous system metastases (CNS) and/or cancerous meningitis;
9. Any component of a product or preparation similar to the study drug PD-1 monoclonal antibody has ever caused a severe allergic reaction, including known severe allergic reaction to other monoclonal antibodies, oxaliplatin, S-1 and other related compounds (NCI-CTCAE V5.0≥3);
10. a known history of hereditary bleeding or a blood clotting disorder that is at risk of bleeding;
11. Patients who underwent major surgery within 4 weeks;
12. Subjects who did not recover from complications from previous surgery, i.e., did not drop to ≤1 (CTCAE version 5.0) (excluding hair loss and fatigue);
13. Immunosuppressive drugs should be used for 2 weeks or within 2 weeks or during the study, excluding the following situations:

    A) Intranasal, inhaled, topical or topical steroid injections (e.g. intraarticular); B) Systemic corticosteroids at physiological dose (≤10mg/day prednisone or equivalent); C) short-term (≤7 days) use of steroids to prevent or treat non-autoimmune allergic diseases;
14. Subjects with active or preexisting autoimmune diseases that are likely to recur;
15. Subjects with a known history of idiopathic pulmonary fibrosis, drug-induced pneumonia, histological pneumonia, or non-infectious pneumonia;
16. known active tuberculosis history;
17. A history of human immunodeficiency virus infection (HIV positive), other acquired or congenital immunodeficiency diseases, or a history of organ transplantation, or stem cell transplantation;
18. The hepatitis B or C virology test meets any of the following criteria at the time of screening:

    A) HBsAg positive, and the titer of HBV-DNA in peripheral blood ≥104 copy number /mL or ≥2000IU/mL (HBV carriers should be treated with antiviral therapy by the researcher as appropriate); B) Active hepatitis C: HCV antibody positive and HCV-RNA higher than the detection limit of the analytical method;
19. Subjects had active or uncontrollable infections requiring systematic treatment within 2 weeks before randomization;
20. have received live virus vaccine within 4 weeks;
21. The presence of uncontrollable pleural effusion, pericardial effusion or ascites requiring repeated drainage or medical intervention;
22. gastrointestinal perforation and/or fistula occurred within 6 months, and gastrointestinal bleeding of clinical significance occurred within 3 months before randomization;
23. have intestinal obstruction or the following diseases or history: inflammatory bowel disease or general bowel resection (partial colon resection or general small bowel resection with chronic diarrhea), Crohn's disease, ulcerative colitis or chronic diarrhea;
24. with severe medical problems, such as level III and above abnormal cardiac function (NYHA), ischemic heart disease (such as myocardial infarction, or angina pectoris) such as cardiovascular disease, or a history of myocardial infarction , within 3 months after the drug of poorly controlled diabetes (FPG)≥10mmol/L) or poorly controlled hypertension, systolic blood pressure≥160mmHg and/or diastolic blood pressure≥100mmHg;
25. Subjects who are lactating or who plan to become pregnant during treatment and within 6 months after treatment;
26. subjects who are unwilling to receive effective contraceptives during treatment and within 6 months after treatment (including male subjects who are capable of making a woman pregnant and female subjects and their male partners);
27. The investigator believes that subjects are not suitable for the study because of other conditions that may affect their compliance with the protocol and evaluation of the study indicators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
pathologic complete response (PCR) | 6month
  The enhancement lesions disappeared completely

SECONDARY OUTCOMES:
R0 resection rate | 6month
  R0 resection rate
ORR | 12month
  Objective response rate
Percentage of Progression-free survival (1-PFSR) | 12month
  Percentage of Progression-free survival of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Chengxue Dang, PhD, Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- The First Affiliated Hospital of Xi 'an Jiaotong University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No